CLINICAL TRIAL: NCT04488731
Title: The Effect of Coffee Consumption and Body Weight on the Serum Levels of Leptin, Folic Acid, and Vitamin B12 in Young Males: A Cross-Sectional Study
Brief Title: The Effect of Coffee Consumption on the Serum Levels of Leptin, Folic Acid, and Vitamin B12
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-PHA-19
Record Dates: First submitted 2020-07-19; First posted 2020-07-28 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Atherosclerosis
Keywords: Coffee; BMI; Leptin; Folic acid; Vitamin B12
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples will be retained
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NW/MCC: Normal body mass index (BMI) / with moderate coffee consumption
  Interventions: Behavioral: Normal BMI and moderate coffee consumption
- NW/HCC: Normal body mass index (BMI) / with heavy coffee consumption
  Interventions: Behavioral: Normal BMI and heavy coffee consumption
- OW/MCC: Overweight / with moderate coffee consumption
  Interventions: Behavioral: overweight and moderate coffee consumption
- OW/HCC: Overweight / with heavy coffee consumption
  Interventions: Behavioral: overweight and heavy coffee consumption

INTERVENTIONS:
Behavioral: Normal BMI and moderate coffee consumption — Normal BMI and moderate coffee consumption
  Groups: NW/MCC
Behavioral: Normal BMI and heavy coffee consumption — Normal BMI and heavy coffee consumption
  Groups: NW/HCC
Behavioral: overweight and moderate coffee consumption — overweight and moderate coffee consumption
  Groups: OW/MCC
Behavioral: overweight and heavy coffee consumption — overweight and heavy coffee consumption
  Groups: OW/HCC

SUMMARY:
The effect of coffee and body weight during the last 3 months on the level of leptin, folic acid, and vitamin B12

DETAILED DESCRIPTION:
Coffee consumption has been associated with several risk factors leading to cardiovascular diseases (CVDs), including hyperhomocysteinemia and hyperlipidemia. Frequent coffee consumption has beneficial effects in reducing the risk of diabetes mellitus (DM) type 2, obesity, liver disease, CVDs, some types of cancer, Parkinson's disease, and Alzheimer's disease. Controversies concerning coffee consumption benefits and risks in regards for CVDs were mentioned in many studies. Folic acid and vitamin B12 are necessary vitamins in homocysteine metabolism which is a risk factor for atherosclerosis. Leptin, is a hormone linked to obesity and it could be related to atherosclerosis.

The combined effect of coffee consumption and body weight on the levels of leptin, folic aid, and vitamin B12 is not well studied. In our study, we will study the effect of coffee consumption in males with different body mass indices to see the effect of several important parameters such as leptin, Folic acid, and vitamin B12.

ELIGIBILITY:
Inclusion Criteria:

* male,
* ASU student,
* do not have any acute or chronic medical conditions.

Exclusion Criteria:

* students who used any medications for either an acute and/or a chronic condition during the past 3 months prior to the study entry.

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only young males are considered
Study Population: Young male students studying at Applied Science Private University (ASU) in Amman were approached for study participation.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-07-26 (Actual); Primary Completion 2020-09-26 (Estimated); Study Completion 2020-10-26 (Estimated)

PRIMARY OUTCOMES:
leptin | Baseline
  Plasma Concentration of leptin in ng /ml
folic acid | Baseline
  Plasma Concentration of folic acid in ng /ml
Vitamin B12 | Baseline
  Plasma Concentration of Vitamin B12 in pg /ml

SECONDARY OUTCOMES:
fasting blood glucose | Baseline
  Plasma Concentration of glucose mg/dL
lipid profile | Baseline
  Plasma Concentration of LDL, HDL in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-samak, PhD, Principal Investigator — Applied Sciences Private University
Locations (1):
- Applied Science University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underline results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published
Access Criteria: Open access

REFERENCES:
- [Result] Grubben MJ, Boers GH, Blom HJ, Broekhuizen R, de Jong R, van Rijt L, de Ruijter E, Swinkels DW, Nagengast FM, Katan MB. Unfiltered coffee increases plasma homocysteine concentrations in healthy volunteers: a randomized trial. Am J Clin Nutr. 2000 Feb;71(2):480-4. doi: 10.1093/ajcn/71.2.480. PMID 10648261
- [Result] Ma Y, Peng D, Liu C, Huang C, Luo J. Serum high concentrations of homocysteine and low levels of folic acid and vitamin B12 are significantly correlated with the categories of coronary artery diseases. BMC Cardiovasc Disord. 2017 Jan 21;17(1):37. doi: 10.1186/s12872-017-0475-8. PMID 28109191
- [Derived] Hasoun LZ, Khader HA, Abu-Taha MI, Mohammad BA, Abu-Samak MS. A Cross-Sectional Study on the Combined Effect of Body Weight and Coffee Consumption on Serum Levels of Leptin, Vitamin B12, and Folic Acid in Healthy Young Adult Males. J Multidiscip Healthc. 2021 Mar 15;14:639-650. doi: 10.2147/JMDH.S290990. eCollection 2021. PMID 33758508